CLINICAL TRIAL: NCT02804061
Title: Strategizing the Best Approach to Prevent Early Excessive Gestational Weight Gain Using a Nutrition and Exercise Lifestyle Intervention Program (NELIP)
Brief Title: Early Prevention of Excessive Gestational Weight Gain Using Lifestyle Change
Acronym: NELIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Iowa State University (Other)
Responsible Party: Principal Investigator, Michelle Mottola, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 108080
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Excessive Weight Gain in Pregnancy, First Trimester; Excessive Weight Gain in Pregnancy With Baby Delivered; Birth Weight
Keywords: nutrition; exercise; behavior change; adherence
MeSH Terms: conditions — Birth Weight; Motor Activity | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full NELIP (Active Comparator): This group will receive the full Nutrition and Exercise Lifestyle Intervention Program (two behavior changes) from enrollment until birth and serves as the comparator control (Group A).
  Interventions: Behavioral: NELIP
- Nutrition followed by Exercise (N+E) (Experimental): Intervention - Nutrition component only (one behaviour) until 24 week assessment, then the addition of the second behavior change (Exercise component) at 25 weeks, with both behaviours followed until birth (Group B).
  Interventions: Behavioral: NELIP
- Exercise followed by Nutrition (E+N) (Experimental): Intervention - Exercise component only (one behaviour) until 24 week assessment, after which there will be the addition of the second behaviour change (Nutrition component), with both behaviours followed until birth (Group C).
  Interventions: Behavioral: NELIP

INTERVENTIONS:
Behavioral: NELIP
  Other Names: Nutrition and Exercise Lifestyle Intervention Program

SUMMARY:
Nutrition and exercise behaviour change programs can prevent excessive gestational weight gain (EGWG). The Nutrition and Exercise Lifestyle Intervention Program (NELIP) is a previously published two-behaviour change program which was successful in preventing EGWG across normal weight, overweight and obese pre-pregnancy body mass index (BMI) categories (Ruchat et al. 2012; Mottola et al. 2010), however some women found it difficult to adhere to two lifestyle behaviour changes throughout pregnancy. The proposed pilot randomized controlled trial will address the issue of adherence by identifying the best way to offer a two-behaviour change program (NELIP) to pregnant women to increase the effectiveness of preventing early and total EGWG. Participants will begin the program at <18 weeks gestation and will be randomized to one of three groups: A) Receive both behaviour changes (Nutrition AND Exercise) simultaneously at entrance to the study; B) Receive the nutrition component first followed sequentially by the introduction of exercise at 25 weeks gestation (Nutrition FOLLOWED by Exercise); C) Receive the exercise component first followed sequentially by the introduction of the nutrition component at 25 weeks gestation (Exercise FOLLOWED by Nutrition).

DETAILED DESCRIPTION:
A randomized parallel groups design will be used as a pilot project. Each participant will be medically pre-screened using the PARmed-X for Pregnancy (2015) in early pregnancy (<18 weeks), stratified by pre-pregnancy BMI status (normal weight [18.5-24.9 kg/m2]; overweight [25.0-29.9 kg/m2], obese [=>30.0 kg/m2]) and randomized into one of 3 groups: Group A) NELIP (full intervention); Group B) Nutrition intervention given at study entry followed sequentially by the exercise intervention starting immediately after 24 week mid-way visit (N+E); or Group C) Exercise intervention started at study entry followed sequentially by the nutrition intervention starting immediately after 24 week mid-way visit (E+N). Infant sex, body weight, length, complications will be recorded at birth and the last known maternal body weight. Neonatal morphometrics will be assessed with diaper only (6 skinfold sites from umbilical, suprailiac, biceps, triceps, subscapular, and anterior thigh; circumferences from the head, chest, abdomen, hips, thigh, leg, arm, and arm, forearm, thigh and leg length measured to the nearest mm) and will be measured within 6-18 hours of delivery by a member of the research team visiting the woman either at hospital or home. Each maternal-infant pair will be asked to return to the lab at 2, 6 and 12 months post-delivery for follow-up and assessment of chronic disease risk.

ELIGIBILITY:
Inclusion Criteria:

* single pregnancy (no twins);
* < 18 weeks, 0 days pregnant at time of entry to study;
* low-risk pregnancy, as determined by medical pre-screening via PARmed-X for Pregnancy by their health care provider;
* > 18 years of age;
* low physical activity defined as less than 3 intentional bouts of 30 minutes of moderately intense physical activity per week;
* non smokers.

Exclusion Criteria:

* multiple pregnancy (twins, etc);
* contraindication to exercise (includes chronic diseases such as cardiovascular diseases, thyroid diseases, uncontrolled Type 2 diabetes, peripheral vascular disease, hypertension);
* > 18 weeks, 0 days pregnant at time of entrance to study;
* <18 years of age;
* high physical activity defined as more than 3 intentional bouts of 30 minutes of moderately intense physical activity per week;
* smokers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Prevention of early excessive gestational weight gain | Up to 24 weeks gestation
  Calculations based on the Institute of Medicine (2009) weight gain guidelines

SECONDARY OUTCOMES:
Prevention of total excessive gestational weight gain | Up to 38 weeks of pregnancy or last known pregnancy weight
  Calculations based on the Institute of Medicine (2009)
Birth weight | At Birth
  Taken from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F Mottola, PhD, Principal Investigator — Western University, Canada
Locations (1):
- Exercise and Pregnancy Lab, 2245, 3-M Centre - University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruchat SM, Davenport MH, Giroux I, Hillier M, Batada A, Sopper MM, Hammond JM, Mottola MF. Nutrition and exercise reduce excessive weight gain in normal-weight pregnant women. Med Sci Sports Exerc. 2012 Aug;44(8):1419-26. doi: 10.1249/MSS.0b013e31825365f1. PMID 22453250
- [Background] Mottola MF, Giroux I, Gratton R, Hammond JA, Hanley A, Harris S, McManus R, Davenport MH, Sopper MM. Nutrition and exercise prevent excess weight gain in overweight pregnant women. Med Sci Sports Exerc. 2010 Feb;42(2):265-72. doi: 10.1249/MSS.0b013e3181b5419a. PMID 20083959
- [Background] Davenport MH, Ruchat SM, Giroux I, Sopper MM, Mottola MF. Timing of excessive pregnancy-related weight gain and offspring adiposity at birth. Obstet Gynecol. 2013 Aug;122(2 Pt 1):255-261. doi: 10.1097/AOG.0b013e31829a3b86. PMID 23969792
- [Result] Nagpal TS, Prapavessis H, Campbell C, Mottola MF. Measuring Adherence to a Nutrition and Exercise Lifestyle Intervention: Is Program Adherence Related to Excessive Gestational Weight Gain? Behav Anal Pract. 2017 May 17;10(4):347-354. doi: 10.1007/s40617-017-0189-5. eCollection 2017 Dec. PMID 29214130
- [Result] Nagpal TS, Prapavessis H, Campbell CG, de Vrijer B, Bgeginski R, Hosein K, Paplinskie S, Manley M, Mottola MF. Sequential Introduction of Exercise First Followed by Nutrition Improves Program Adherence During Pregnancy: a Randomized Controlled Trial. Int J Behav Med. 2020 Feb;27(1):108-118. doi: 10.1007/s12529-019-09840-0. PMID 31872340
- [Derived] Bgeginski R, Nagpal TS, Hosein K, Manley M, Paplinskie S, Prapavessis H, Campbell CG, DE Vrijer B, Mottola MF. Does Delivery of a Nutrition and Exercise Intervention Simultaneously or Sequentially Prevent Excessive Gestational Weight Gain? The NELIP Trial. Med Sci Sports Exerc. 2025 Sep 1;57(9):2032-2039. doi: 10.1249/MSS.0000000000003729. Epub 2025 Apr 8. PMID 40197635